CLINICAL TRIAL: NCT05388435
Title: A Phase 1/2, Open-Label, Multicenter, Dose-Finding Study of SKL27969 to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy in Patients With Advanced Solid Tumors
Brief Title: Safety, Tolerability, PK/PD & Preliminary Efficacy of SKL27969 in Advanced Solid Tumors Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study has been terminated based on portfolio prioritization. No safety trends or issues were identified at any dose level.
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SKL27969C001
Record Dates: First submitted 2022-03-15; First posted 2022-05-24 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Malignant Solid Tumors; Glioblastoma; Non-Small Cell Lung Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Glioblastoma; Carcinoma, Non-Small-Cell Lung; Triple Negative Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Part 1, Phase 1 Dose Escalation and Part 2, Phase 2 Dose Expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation Phase (Experimental): Part 1 is a dose escalation phase to evaluate the safety, tolerability, and define the MTD and RP2D. Part 1 is a 3+3 design.
  Interventions: Drug: SKL27969
- Part 2: Dose Expansion Phase (Experimental): Part 2 includes tumor-specific expansion cohorts utilizing the MTD/RP2D doses (determined from Part 1) to further explore safety and anti-tumor activity of SKL27969, in addition to the PK and PD from the patients with the selected tumor types.
  Interventions: Drug: SKL27969

INTERVENTIONS:
Drug: SKL27969 — SKL27969 will be orally administered once daily on an intermittent dosing schedule (3 days on and 4 days off).

SUMMARY:
Primary Objective of Part 1 (Dose Escalation Phase): Evaluate the safety and tolerability of SKL27969, and determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of SKL27969

Primary Objective of Part 2 (Dose Expansion Phase): Evaluate the preliminary anti-tumor activity of SKL27969

DETAILED DESCRIPTION:
Secondary Objectives of Part 1 (Dose Escalation Phase):

1. Characterize the pharmacokinetic (PK) profile of SKL27969
2. Evaluate the preliminary anti-tumor activity of SKL27969

Secondary Objectives of Part 2 (Dose Expansion Phase):

1. Investigate the safety and tolerability of SKL27969 at the RP2D in patients with selected tumor types
2. Characterize the PK of SKL27969

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written, voluntary informed consent prior to any study-specific procedures;
2. Male and female patients at least 18 years of age at the time of informed consent;
3. Histologically or cytologically confirmed diagnosis of non-resectable or metastatic solid malignancy that is refractory (radiographic documentation of progression) or intolerant of established therapies known to provide clinical benefit for the malignancy in the opinion of the Investigator;
4. Evidence of radiological progressive disease and minimum life expectancy of at least months, in the judgement of the Investigator;
5. Measurable disease per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1 or Response Assessment in Neuro-Oncology (RANO), with the last imaging performed within 28 days before Cycle 1 Day 1, and documented disease progression during or after their most recent line of anticancer therapy;
6. 6. Prior treatment required for the following diagnoses that are histologically and molecularly confirmed:

   1. Recurrent high-grade glioma (HGG) (e.g., anaplastic astrocytoma (high grade), recurrent ependymoma BRAFV600E or GBM) must have biopsy proven evidence according to 2021 World Health Organization (WHO) classification (Grade 3 or 4) and received:

      - Radiotherapy with at least 2 cycles of temozolomide chemotherapy
   2. NSCLC of any histologic sub-type with local mutational analysis; must have received platinum-based therapy, immune checkpoint inhibitor and targeted tyrosine kinase inhibitor, if mutation present for approved agent in accordance with product labels; or
   3. TNBC must have biopsy proven evidence according to the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines and received

      * Checkpoint inhibitors for patients who are PD-L1 positive;
      * PARP inhibitors for patients with germline BRCA mutations; or
      * Targeted antibody-drug conjugates, such as Sacituzumab govitecan.
7. Must have recovered to Grade 1 from the effects of any prior investigational systemic therapies; with the exception of alopecia and Grade 2 peripheral neuropathy;
8. Recurrent HGG must be neurologically stable for 7 or more days and takes no more than 2 mg or 4 mg of dexamethasone or equivalent steroid per day;
9. ECOG performance status of 0 or 1;
10. Willing to follow the contraception requirements as outlined (refer to Section 13.2 for details):

    a. For Women:

    Women of childbearing potential:
    * Negative pregnancy test;
    * Compliant with at least 2 effective contraceptive methods (e.g., oral contraceptives, condom with spermicide, etc) used at the same time during the study and for 90 days after the last dose of study drug; and
    * Abstinence is not considered an adequate contraceptive method.

    Women of non-childbearing potential:
    * Must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy) or postmenopausal (defined as no menstrual cycle for at least 12 consecutive months). b. For Men:
    * Must be surgically sterile, or compliant with a contraceptive method (effective barrier contraception, such as condom with spermicide) during the study and for 90 days from the last dose of study drug.

    Male patients with female partner(s) of childbearing potential:
    * Female partner must use a highly effective methods of contraception (e.g., oral contraceptives, etc). Male patients with female partner(s) of non-childbearing potential (i.e., postmenopausal or surgically sterile for at least 6 months prior to Screening):
    * No additional contraception method is required.
11. Hematological and biochemical indices within the ranges shown below:

    1. Hemoglobin equal to or more than 9 g/dL (transfusion to achieve this is allowed);
    2. Neutrophils equal to or more than 1.5 X 10 degree/L; and
    3. Platelet count equal to or more than100 X 109 degree/L (transfusion to achieve this is allowed).
12. Hepatic function: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) less than or equal to 1.5 X upper limit of normal (ULN), patient with liver metastases less than or equal to 5 X ULN, and serum bilirubin less than or equal to 1.5 X ULN;
13. Renal function: Creatinine clearance greater than or equal to 45 mL/min as determined by Cockcroft-Gault;
14. Cardiac function criteria: Left ventricular ejection fraction of greater than or equal to 50% as assessed by multi-gated acquisition or ultrasound/echocardiography; corrected QT interval less than or equal to 470 ms;
15. Consent to appropriate protection from direct sunlight (e.g., utilizing sunscreen daily, protective clothing, UV protection sunglasses), and avoid artificial tanning during the study participation;
16. Able to swallow oral medication; and
17. Willing and able to comply with all protocol required visits and assessments.

Exclusion Criteria:

1. Patient has had 1 or more of the following cardiac function criteria:

   1. Clinically meaningful unstable angina;
   2. Myocardial infarction within 6 months prior to starting the study treatment;
   3. New York Heart Association Class II or greater congestive heart failure;
   4. QT interval corrected using Fridericia's formula >470 msec obtained as the mean from 3 consecutive resting ECGs;
   5. Clinically significant abnormalities in rhythm, conduction, or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block);
   6. Ongoing congestive heart failure or cardiac dysrhythmias of National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) greater than or equal to Grade 2 or uncontrolled atrial fibrillation;
   7. Congenital long QT syndrome;
   8. Cerebrovascular accident within 6 months prior to starting the study treatment; or
   9. Clinically significant arterial hypertension despite medical treatment.
2. Female patient is pregnant, breast-feeding, intending to donate ova, or planning to become pregnant before, during or within at least 90 days after the final study drug administration;
3. Male patient intends to father or donate sperm during the study or for at least 90 days after the final study drug administration;
4. History of major gastrointestinal surgery, inflammation, or condition that can impair absorption of study drug;
5. Evidence of infections (including chronic hepatitis type B or C and human immunodeficiency virus (HIV) infection, if status known);
6. Active infection requiring intravenous (IV) antibiotics;
7. Prior participation in another clinical study with PRMT5 inhibitor(s);
8. Known allergies, hypersensitivity or intolerance to PRMT5 inhibitors or SKL27969 and any of its excipients;
9. Requirement of pharmacologic doses of glucocorticoids (e.g., greater than or equal to 10 mg of prednisone) with the exception of patients diagnosed with glioma;
10. Any unstable or severe ongoing medical/psychiatric conditions, as well as medical history, laboratory, imaging, ECG, or other clinically important findings that, in the opinion of the Investigator, can indicate an unacceptable risk for the patient's participation in the study;
11. Received any systemic anti-cancer therapy including but not limited to chemotherapy, targeted agents, antibody therapy for cancer, immunotherapy for cancer, hormonal therapy, or an investigational agent within 4 weeks prior to start of study drug treatment;
12. Active secondary malignancy within 3 years except basal or squamous cell carcinoma;
13. Major surgery within 4 weeks prior to start of study drug treatment;
14. Radiation therapy within 4 weeks prior to start of study drug treatment (palliative radiation or stereotactic radiosurgery within 7 days prior to start of the study drug treatment). Patients must have recovered from all acute radiotherapy-related toxicities;
15. History of alcohol or drug abuse for the past 5 years;
16. Patients must not use proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole, pantoprazole, etc) at least 7 days prior to the first dose of SKL27969 and throughout the study; or
17. Concurrent therapy with drugs known to be potent (strong or moderate) inhibitors and inducers of cytochrome P450(CYP)3A4, including grapefruit, grapefruit juice, or grapefruit-containing products and grapefruit-related citrus fruits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Part 1 (Dose Escalation Phase) - Numbers of participants with adverse events, dose interruptions and modifications | 1 year
  Any incidence of AEs, dose interruptions and dose modifications from signing of Informed Consent Form (ICF) until discontinuation and/or protocol required Survival Follow-up is completed.
Part 1 (Dose Escalation Phase) - Number of participants with dose limiting toxicities | 1 year
  The Dose Limiting Toxicities (DLTs) are based on drug related adverse events and defined as any of the following events: hematological / non-hematological toxicity of Grade 3 or higher.
Part 1 (Dose Escalation Phase) - Number of participants with abnormal assessments | 1 year
  Post baselines changes in laboratory assessments, vital signs, electrocardiograms (ECGs) and physical examinations related to SKL27969.
Part 2 (Dose Expansion Phase) - Number of participants with partial response data | 30 months
  ORR is defined as the proportion of participants who have a partial response (PR) or better according to the RECIST version 1.1 or RANO.
Part 2 (Dose Expansion Phase) - Number of participants with progression-free survival | 30 months
  Each participant will be assessed for progression-free survival (PFS) starting from first day of treatment until disease progression according to RECIST version 1.1 or RANO.
Part 2 (Dose Expansion Phase) - Number of participants with overall survival | 30 months
  Each participant will be assessed for overall survival (OS) starting from first day of treatment until death.

SECONDARY OUTCOMES:
Part 1 (Dose Escalation Phase) - Number of participants with partial response data | 1 year
  ORR is defined as the proportion of participants who have a partial response (PR) or better according to the RECIST version 1.1 or RANO.
Part 2 (Dose Expansion Phase) - Number of participants with adverse events, dose interruptions and modifications | 30 months
  Any incidence of AEs, dose interruptions and dose modifications from signing of Informed Consent Form (ICF) until discontinuation and/or protocol required Survival Follow-up is completed.
Part 2 (Dose Expansion Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for Cmax
Part 2 (Dose Expansion Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for AUC∞
Part 2 (Dose Expansion Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for AUC0-t
Part 2 (Dose Expansion Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for AUC0-tau
Part 2 (Dose Expansion Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for tmax
Part 2 (Dose Expansion Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for t½
Part 2 (Dose Expansion Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for CL/F
Part 2 (Dose Expansion Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for accumulation ratio (AR)
Part 1 (Dose Escalation Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for Cmax
Part 1 (Dose Escalation Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated AUC∞
Part 1 (Dose Escalation Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for AUC0-t
Part 1 (Dose Escalation Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for AUC0-tau
Part 1 (Dose Escalation Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for tmax
Part 1 (Dose Escalation Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for t½
Part 1 (Dose Escalation Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for CL/F
Part 1 (Dose Escalation Phase) - Pharmacokinetics of SKL27969 | 30 months
  Will be calculated for accumulation ratio (AR)

CONTACTS AND LOCATIONS:
Overall Officials: Vijaykumar Vashi, PhD, Study Chair — SK Life Science, Inc.
Locations (4):
- United States (4):
  - City of Hope, Duarte, California
  - START Midwest, Grand Rapids, Michigan
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - MD Anderson Cancer Center, Houston, Texas